CLINICAL TRIAL: NCT06847503
Title: Functional Outcome After Combined Posterior Laminectomy and Anterior Cervical Discectomy and Fusion for Large Cervical Disc Prolapse
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrahman Zakaria Abdelrahman, residant doctor, Assiut University
Other Study IDs: Post Laminectomy Ant Cervical
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cervical Disc Prolapse
Keywords: Posterior Laminectomy; Anterior Cervical Discectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group A: Patients with degenerative large cervical disc prolapse and canal stenosis with myelopathy.
  (we defined large cervical disc prolapse as any cervical disc prolapse occupying 40% or more of the cervical spinal canal)

SUMMARY:
Cervical disc herniation (CDH) is the result of the displacement of the nucleus pulposus of the intervertebral disc, which may result in impingement of the traversing nerves as they exit the neural foramen or directly compressing the spinal cord contained within the spinal canal.[1] Eventually symptoms may arise because of a CDH with compression of the rootlet or spinal cord.[2] When conservative treatment for CDH fails, surgical treatment may be considered.[3] The main goals of surgical treatment are to remove pressure from the nerves, restore the alignment of the vertebrae, to stabilize the spine [3] and to prevent progression of neurological deficit in case of myelopathy.[4] Anterior cervical discectomy and fusion (ACDF) has proven to be an effective surgical intervention for both cervical radiculopathy and myelopathy and has become standard treatment for both of these disease states over the last half-century.[5] Certain reports have indicated that various complications are associated with ACDF namely, incomplete decompression, recurrence of myelopathy due to adjacent segment degeneration.[6] In cases where the stenosis is extensive, or attributed in part to congenital stenosis, the posterior approach may be advantageous to achieve more extensive decompression that would otherwise not be possible through an anterior approach.[7] Given that most stenosis occurs from anterior pathology, a posterior decompression works to indirectly relieve pressure on the spinal cord.[8] Misalignment and large anterior compression of the spinal cord can be risk factors for insufficient functional recovery in patients treated with posterior decompression alone.[9] In a study of 428 patients that were enrolled in a prospective cohort study to investigate the incidence, etiology, and outcomes of patients who experience neurological deterioration after surgery for degenerative cervical myelopathy(DCM), Evaniew et al[10] reported the incidence of deterioration after surgery for DCM was approximately one in ten (12%).

In this study we will perform combined posterior laminectomy and ACDF to avoid incomplete decompression and neurological deterioration after surgery. We aim to assess the functional outcome after combined posterior laminectomy and ACDF in patients with large cervical disc prolapse.

In this study we will perform combined posterior laminectomy and ACDF to avoid incomplete decompression and neurological deterioration after surgery. We aim to assess the functional outcome after combined posterior laminectomy and ACDF in patients with large cervical disc prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative large cervical disc prolapse and canal stenosis with myelopathy.

(we defined large cervical disc prolapse as any cervical disc prolapse occupying 40% or more of the cervical spinal canal)

Exclusion Criteria:

* Cervical disc prolapse with wide canal
* Cervical disc prolapse with radiculopathy
* Traumatic Cervical disc prolapse
* Patients with ossification of the posterior longitudinal ligament (OPLL)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with degenerative large cervical disc prolapse and canal stenosis with myelopathy.
  (we defined large cervical disc prolapse as any cervical disc prolapse occupying 40% or more of the cervical spinal canal)
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement in the modified Japanese Orthopaedic AssociationmJOA-AR scale. | 30 day
  It is an 18-point scale that addresses upper (5 points) and lower extremity (7 points) motor function, sensation (3 points) and micturition (3 points). A score of 18 reflects no neurological deficits whereas a lower score indicates a greater degree of disability and functional impairment. The mJOA is the second most commonly used outcome measure to quantify severity in patients with DCM